CLINICAL TRIAL: NCT04844060
Title: Analysis of Clinical Data and Diagnosis in Any Person Requiring an Assay of Alzheimer Biomarkers in Cerebrospinal Fluid
Brief Title: Cerebro Spinal Fluid Collection (CSF)
Acronym: Analzheimer
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: DC-2009-1002
Record Dates: First submitted 2021-03-29; First posted 2021-04-14 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Alzheimer Disease; Dementia With Lewy Bodies; Frontotemporal Dementia; Parkinson's Disease Dementia; Multiple System Atrophy
Keywords: CSF library; Database of patients with cognitive disorders
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Frontotemporal Dementia; Multiple System Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cognitive impairment: All patients with cognitive disorders observed at the memory center of Strasbourg and in whom a lumbar puncture is performed as part of the patient's diagnosis.
  Interventions: Other: Lumbar punction

INTERVENTIONS:
Other: Lumbar punction — Lumbar punction

SUMMARY:
Cognitive neurodegenerative diseases are a major public health issue. At present, the diagnosis of certainty is still based on anatomopathological analyses. Even if the diagnostic tools available to clinicians have made it possible to improve probabilistic diagnosis during the patient's lifetime, there are still too many diagnostic errors and sub-diagnostic in this field. The arrival of biomarkers has made it possible to reduce these diagnostic errors, which were of the order of 25 to 30%. This high error rate is due to different parameters. These diseases are numerous and often present common symptoms due to the fact that common brain structures are affected. These diseases evolve progressively over several years and their early diagnosis, when the symptoms are discrete, makes them even more difficult to diagnose at this stage. In addition, co-morbidities are common in the elderly, further complicating the diagnosis of these diseases.

At present, the only cerebrospinal fluid (CSF) biomarkers that are routinely used for the biological diagnosis of neurodegenerative cognitive pathologies are those specific to Alzheimer's disease: Aβ42, Aβ40, Tau-total and Phospho-Tau. These biomarkers represent an almost indispensable tool in the diagnosis of dementia.

It is therefore important to determine whether Alzheimer's biomarkers can be disrupted in other neurodegenerative cognitive pathologies, but also to find biomarkers specific to these different pathologies by facilitating the implementation of clinical studies which will thus make it possible to improve their diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lumbar puncture (LP)
* Patients with accurate clinical diagnosis

Exclusion Criteria:

* Patients who do not have a lumbar puncture
* Patients for whom no accurate diagnostic information is available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with cognitive disorders observed at the memory center of Strasbourg and in whom a lumbar puncture is performed as part of the patient's diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-02 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
CSF collection | 1 year
  To create a database of patients with cognitive disorders in whom a lumbar puncture has been carried out in order to measure Alzheimer's biomarkers. This database would not only be biological but also clinical and diagnostic, including the results of neuropsychological tests, clinical examinations, the results of brain imaging (MRI, PET-FDG, DAT-SCAN,…) as well as the last diagnosis retained by the clinician in charge of the patient. Thus, after completing this database, the main objective is to evaluate the proportion of different diseases that have led to the decision to search for Alzheimer biomarkers in CSF.

SECONDARY OUTCOMES:
Setting up in new study/collaboration | 1 year
  This database would allow clinical studies and collaborations to be built easily and quickly.
  For example, when setting up a clinical study with the aim of testing the discriminating potential of a biomarker between various cognitive pathologies, we will only use in this database patients for whom the diagnosis is well established. The objective will be to determine whether the biomarker is capable of discriminating between these well-defined populations.

OTHER OUTCOMES:
To compare the levels of CSF Alzheimer's biomarkers between these different populations and determine their ability to discriminate between AD and other neurodegenerative cognitive pathologies | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric BLANC, MD/PhD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service d'évaluation et Centre Mémoire de Ressources et de Recherche (CM2R), Hôpital de jour Saint François - Pôle de Gériatrie, Hôpitaux Universitaires de Strasbourg, Hôpital de la Robertsau, Strasbourg, France